CLINICAL TRIAL: NCT02588378
Title: In Vivo Visualization of Active Macrophages and Retinal Pigment Epithelium (RPE) Damage in Age Related Macular Degeneration (AMD) & Related Conditions
Brief Title: The Role of Inflammation in AMD and Related Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 15-052
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (9):
- Early dry AMD (no GA): multi-modal cSLO imaging
  Interventions: Procedure: multi-modal cSLO imaging
- Late dry AMD (with GA): multi-modal cSLO imaging
  Interventions: Procedure: multi-modal cSLO imaging
- Reticular Pseudodrusen (RPD): multi-modal cSLO imaging
  Interventions: Procedure: multi-modal cSLO imaging
- Polypoidal Choroidal Vasculopathy (PCV): multi-modal cSLO imaging
  Interventions: Procedure: multi-modal cSLO imaging
- Retinal Angiomatous Proliferaion (RAP): multi-modal cSLO imaging
  Interventions: Procedure: multi-modal cSLO imaging
- Central Serous Retinopathy (CSR): multi-modal cSLO imaging
  Interventions: Procedure: multi-modal cSLO imaging
- RPE Detachment (RPED): multi-modal cSLO imaging
  Interventions: Procedure: multi-modal cSLO imaging
- New onset CNVM (wet AMD): multi-modal cSLO imaging
  Interventions: Procedure: multi-modal cSLO imaging
- Healthy (non-AMD) controls: multi-modal cSLO imaging
  Interventions: Procedure: multi-modal cSLO imaging

INTERVENTIONS:
Procedure: multi-modal cSLO imaging

SUMMARY:
This prospective, non-therapeutic study will compare the relative utility of multiple ocular imaging modalities in the detection of the cellular immune response in patients with AMD and related disorders.

ELIGIBILITY:
Inclusion Criteria STUDY EYE

Any tentative clinical diagnosis of the following:

1. Early dry AMD (drusen) with clinical suspicion of CNV
2. Late dry AMD (GA) with clinical suspicion of CNV
3. Reticular Pseudodrusen with clinical suspicion of CNV
4. Polypoidal choroidal vasculopathy
5. Retinal Angiomatous Proliferation
6. Central Serous Retinopathy
7. RPE detachment
8. Conversion to wet AMD (CNV)
9. Decade matched controls

Inclusion Criteria CONTROL EYE

* Subjects > 18 years of age
* Best corrected visual acuity (BCVA) of 20/32 or better

Exclusion Criteria STUDY/CONTROL EYE:

* Patients not able to provide consent for the study.
* Patients with a poor view of the fundus due to cataract or vitreous hemorrhage.
* Patients < 18 years of age
* Patients with known allergy to angiographic dye
* Patients with any concurrent unrelated eye diagnosis that would interfere with image acquisition or interpretation (eg advanced diabetic retinopathy, vascular occlusion, uveitis, or others).

Exclusion Criteria CONTROL EYE

* Suspect diagnosis of AMD, RPD, PCV, RAP, CSR or RPED
* Family history of AMD
* 2 or more large drusen (>125um) or 20 or more medium drusen (64-124um)
* Diabetes
* Patients using Plaquenil/Chloroquine/Hydroxychloroquine
* Diagnosis of inflammatory disease
* Patients with inherited eye disease
* Note: patients with a diagnosis of nevi are NOT excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male or female, 18 years of age or older, able to understand the study protocol and provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-04; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Visualization of RPE damage and presumptive immune cells | 8 months
  Qualitative

CONTACTS AND LOCATIONS:
Overall Officials: Shelley Boyd, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St Michael's Hospital, Toronto, Ontario, Canada